CLINICAL TRIAL: NCT07104838
Title: Efficacy and Safety of Non-intubated Versus Intubated Anesthesia in Thoracoscopic Radical Esophagectomy for Esophageal Cancer: A Prospective Randomized Controlled Trial
Brief Title: Non-intubated Versus Intubated Anesthesia in Thoracoscopic Esophagectomy for Esophageal Cancer
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The First Affiliated Hospital of Guangzhou Medical University (Other)
Responsible Party: Principal Investigator, Jianxing He, head of Guangzhou Institude of respiratory health, The First Affiliated Hospital of Guangzhou Medical University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: EC-TUBELESS-RCT-2025
Record Dates: First submitted 2025-07-29; First posted 2025-08-05 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Esophageal Cancer (EsC)
MeSH Terms: conditions — Esophageal Neoplasms

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intubated (No Intervention)
- Non-intubated (Experimental)
  Interventions: Procedure: Non-intubated spontaneous ventilation anesthesia

INTERVENTIONS:
Procedure: Non-intubated spontaneous ventilation anesthesia — Non-intubated spontaneous ventilation anesthesia
  Arms: Non-intubated

SUMMARY:
This is a prospective, single-center, non-inferiority randomized controlled trial designed to evaluate the perioperative safety and feasibility of non-intubated spontaneous ventilation anesthesia (NIV) compared to conventional intubated mechanical ventilation anesthesia (IMV) in patients undergoing thoracoscopic esophagectomy for esophageal cancer. The study will be conducted at the First Affiliated Hospital of Guangzhou Medical University and aims to assess whether the non-intubated approach can offer comparable or better outcomes in terms of intraoperative and postoperative complications, anesthetic drug consumption, recovery parameters, and overall postoperative rehabilitation.

Eligible patients aged 18 to 75 years with resectable middle or lower thoracic esophageal squamous cell carcinoma or adenocarcinoma (stage I-III) will be randomly assigned (1:1) to receive either NIV using a laryngeal mask airway or IMV with a double-lumen endotracheal tube. Both groups will undergo the same thoracoscopic and laparoscopic surgical procedures, and anesthesia will be managed with standardized protocols. The primary outcome is the incidence of intraoperative and postoperative complications, including hypoxemia, hypercapnia, respiratory failure, and the need for conversion to intubation. Secondary outcomes include anesthetic drug dosage, intraoperative hemodynamic stability, postoperative pain scores, time to ambulation, length of hospital stay, and 30-day readmission rate.

This trial complies with the Declaration of Helsinki. Written informed consent will be obtained from all participants prior to enrollment.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 75 years
* Diagnosed with resectable middle or lower thoracic esophageal squamous cell carcinoma or adenocarcinoma (clinical stage I-III)
* Scheduled to undergo thoracoscopic esophagectomy
* American Society of Anesthesiologists (ASA) score ≤ III
* Eastern Cooperative Oncology Group (ECOG) performance status ≤ 1
* Preoperative pulmonary function test with FEV₁ ≥ 50% predicted
* Written informed consent obtained

Exclusion Criteria:

* Severe risk of aspiration due to reflux, gastric retention, or hiatal hernia
* Body mass index (BMI) ≥ 30 kg/m²
* Extensive pleural adhesions discovered preoperatively
* History of upper thoracic or intrathoracic surgery
* Pregnancy or lactation
* Known allergy or intolerance to anesthetic agents

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of intraoperative and postoperative complications | From anesthesia induction to 30 days postoperatively
  Composite incidence of complications occurring intraoperatively or within 30 days after surgery, including hypoxemia (SpO₂ < 90% for >1 minute), hypercapnia (PaCO₂ ≥ 65 mmHg), conversion to intubation (in the non-intubated group), severe arrhythmia, hemodynamic instability, postoperative pulmonary infection, anastomotic leakage, bleeding, pneumothorax, respiratory failure, and reintubation.